CLINICAL TRIAL: NCT04528511
Title: BurdEn of NEw Onset Atrial FIbrillation in patienTs With Acute Myocardial Infarction: the BENEFIT-AMI Multicenter Prospective Registry
Brief Title: BurdEn of NEw Onset Atrial FIbrillation in patienTs With Acute Myocardial Infarction
Acronym: BENEFIT-AMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Shanghai Tong Ren Hospital (Other); Kaifeng Central Hospital (Other); Shanghai 7th People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Other Study IDs: BENEFIT-AMI
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation New Onset; Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; New-Onset Atrial Fibrillation; Burden; Prospective; Cardiovascular Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low burden of new-onset atrial fibrillation: Patients with MI who are free from a medical history of atrial fibrillation (AF) will be recognized as NOAF if they develop an atrial fibrillation (lasting for at least 30 seconds which are recorded by CEM) incident during hospitalization. Among this subset of patients, those who have a NOAF burden value<10.87% (previously established) will be divided into the low burden group.
  Interventions: Device: Continuous Electronic Monitor
- High burden of new-onset atrial fibrillation: For patients with NOAF complicating AMI, those who have a NOAF burden value≥10.87% (previously established) will be divided into the high burden group.
  Interventions: Device: Continuous Electronic Monitor

INTERVENTIONS:
Device: Continuous Electronic Monitor — All patients with NOAF complicating AMI will receive at least 5 days electronic monitoring for the evaluation of NOAF burden

SUMMARY:
To validate the prognostic importance of the burden of new-onset atrial fibrillation (NOAF) complicating acute myocardial infarction (AMI) in a prospectively designed hospital-based registry. To characterize those factors that contribute to the progression of post-MI NOAF burden. To establish a prediction model for the risk stratification of patients with NOAF complicating AMI. To explore the clinical usefulness of NOAF burden in guiding the anticoagulation therapy among patients with post-MI NOAF.

DETAILED DESCRIPTION:
Our previously designed single-center retrospective cohort study (NCT03533543) suggested that patients with a greater burden of NOAF complicating AMI were challenged by a poor prognosis. In the present study, we aim to design a multicenter, prospective, hospital-based registry to validate the preceding findings. We plan to enroll patients who were admitted for AMI in 9 tertiary medical centers from Shanghai, Henan, and Zhejiang provinces and developed NOAF during the index hospitalization. All eligible patients' demographics, cardiovascular risk factors, comorbidities, laboratory tests, echocardiography data, angiography data, and medications will be collected. NOAF burden is calculated by dividing the total AF duration by the total continuous electronic monitoring (CEM) duration. Other NOAF related characteristics, such as AF pattern, AF frequency, and symptomatic or silent AF, and the longest AF episode duration will also be evaluated. All patients who are discharged alive will be followed for at least 2 years and cardiovascular outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old);
* Patient with AMI (including STEMI and NSTEMI) who developed NOAF during the index hospitalization;
* Patients must have received in-hospital CEM for at least 5 days;
* Patients must give informed consent.

Exclusion Criteria:

* Patients with a medical history of pre-existing AF;
* Patients with a medical history of rheumatic valvular disease;
* Patients with a medical history of sick sinus syndrome;
* Patients undergoing emergent coronary artery bypass surgery;
* Patients who suffer malignant tumors with an expected lifetime less than 1 year ;
* Patients who refuse to receive CEM during hospitalization and the data of heart rhythm cannot be retrieved;
* Patients who refuse to receive percutaneous coronary intervention (PCI) or have contraindications for PCI;
* Patients who have died during the index hospitalization.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with AMI who do not have a medical history of AF and develop an incident AF episode during the index hospitalization.
Sampling Method: Probability Sample
Enrollment: 774 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | up to 1 year
  Death from any cause

SECONDARY OUTCOMES:
Cardiovascular death | up to 1 year
  All deaths without a clear non-cardiovascular cause would be classified as cardiovascular deaths
Heart failure hospitalization | up to 1 year
  Heart failure hospitalization is defined as a minimum of an overnight hospital stay of a participant who presented with symptoms and signs of HF or received intravenous diuretics
Recurrent myocardial infarction | up to 1 year
  Recurrent myocardial infarction is defined as the myocardial infarction episode that occurs after 28 days following the index AMI hospitalization.
Ischemic stroke | up to 1 year
  Ischemic stroke is defined as the presence of a new focal neurologic deficit thought to be ischemic in origin, with signs or symptoms lasting>24h.
Major bleeding | up to 1 year
  Bleeding event with a Bleeding Academic Research Consortium (BRAC) classification of types 3 or 5

CONTACTS AND LOCATIONS:
Overall Officials: Yidong Wei, M.D., Ph.D., Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital
Locations (5):
- China (5):
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Seventh People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tong Ren Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided